CLINICAL TRIAL: NCT05695144
Title: tDCS Combined With rTMS for the Treatment of Negative Symptoms in Patients With Schizophrenia: a Randomized Controlled Trial
Brief Title: tDCS Combined With rTMS for Negative Symptoms of Schizophrenia
Acronym: NIBSNeS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Anding Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Jie Li, Chief physician；professor, Tianjin Anding Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIBSNeS
Record Dates: First submitted 2022-11-15; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Schizophrenia Negative Type
Keywords: rTMS; tDCS; fMRI; ERPs; Cogniton; RCT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS active stimulation combined with rTMS sham stimulation group (Experimental): 1
  Interventions: Device: tDCS active stimulation combined with rTMS sham stimulation
- rTMS active stimulation combined with tDCS sham stimulation group (Experimental): 2
  Interventions: Device: rTMS active stimulation combined with tDCS sham stimulation
- tDCS active stimulation combined with rTMS active stimulation group (Experimental): 3
  Interventions: Device: tDCS active stimulation combined with rTMS active stimulation
- tDCS sham stimulation combined with rTMS sham stimulation group (Experimental): 4
  Interventions: Device: tDCS sham stimulation combined with rTMS sham stimulation

INTERVENTIONS:
Device: tDCS active stimulation combined with rTMS sham stimulation — Active tDCS positive stimulation: left dorsolateral prefrontal cortex (DLPFC) or BeamF3 method; negative stimulation: right frontal, 2mA, 20 mins stimulation, 1 time/day, 5 consecutive days, weekend suspension, lasting 4 weeks, total 20 times.
  Sham stimulation rTMS: Parameters such as stimulation site, current intensity, and stimulation time are kept consistent, keeping the coil facing outward.
  Arms: tDCS active stimulation combined with rTMS sham stimulation group
Device: rTMS active stimulation combined with tDCS sham stimulation — Sham stimulation tDCS: Parameters such as stimulation site, current intensity, and stimulation time are kept consistent, keeping the switch off.
  Active rTMS: stimulation site: left dorsolateral prefrontal cortex (DLPFC); consisting of a total of 3000 pulses per session at 10Hz (4 seconds on and 16 seconds off) at 110% resting motion threshold (RMT), 40 pulses per string; total 75 strings; 1 time/day, 5 consecutive days, weekend suspension, total 20 times. Resting motor thresholds (RMT) were measured before the start of each day of treatment.
  Arms: rTMS active stimulation combined with tDCS sham stimulation group
Device: tDCS active stimulation combined with rTMS active stimulation — Active tDCS positive stimulation: left dorsolateral prefrontal cortex (DLPFC) or BeamF3 method; negative stimulation: right frontal, 2mA, 20 mins stimulation, 1 time/day, 5 consecutive days, weekend suspension, lasting 4 weeks, total 20 times.
  Active rTMS: stimulation site: left dorsolateral prefrontal cortex (DLPFC); consisting of a total of 3000 pulses per session at 10Hz (4 seconds on and 16 seconds off) at 110% resting motion threshold (RMT), 40 pulses per string; total 75 strings; 1 time/day, 5 consecutive days, weekend suspension, total 20 times. Resting motor thresholds (RMT) were measured before the start of each day of treatment.
  Arms: tDCS active stimulation combined with rTMS active stimulation group
Device: tDCS sham stimulation combined with rTMS sham stimulation — Sham stimulation tDCS: Parameters such as stimulation site, current intensity, and stimulation time are kept consistent, keeping the switch off.
  Sham stimulation rTMS: Parameters such as stimulation site, current intensity, and stimulation time are kept consistent, keeping the coil facing outward.
  Arms: tDCS sham stimulation combined with rTMS sham stimulation group

SUMMARY:
Despite major advances in the field of psychopharmacology in recent years, the majority of treated schizophrenia patients retain disabling symptoms, most commonly a variety of negative symptoms. Currently, clinical treatment of schizophrenia remains dominated by pharmacological control. The current use of antipsychotic medications is effective in controlling the positive symptoms of schizophrenia, but has little effect on the negative symptoms. Neuroimaging and neurophysiological studies have shown that negative symptoms are associated with abnormal brain activity in the combined right and left dorsolateral prefrontal and temporoparietal joint regions, and that physical therapy techniques can modulate cortical activity. Therefore, this study aims to investigate the efficacy of transcranial direct current stimulation(tDCS) combined with repetitive transcranial magnetic stimulation(rTMS) on negative symptoms in patients with schizophrenia and to explore possible mechanisms.

The double-blind randomized placebo-controlled study comparing active tDCS stimulation combined with active rTMS stimulation, active rTMS stimulation combined with sham tDCS stimulation, and active tDCS stimulation combined with sham rTMS stimulation to sham tDCS stimulation combined with sham rTMS stimulation at 4 weeks of treatment and 2 weeks of follow-up in patients with predominantly negative symptoms with schizophrenia was studied for efficacy. In addition to the primary observation of changes in the Negative Symptom Assessment Scale (SANS), secondary outcomes include changes in Positive and Negative symptom scale (PANSS) total and negative total scores, changes in the MATRICS Consensus Cognitive Battery (MCCB), changes in local brain activity (functional magnetic resonance imaging, fMRI), white matter integrity (diffusion tensor imaging, DTI), changes in laboratory examination indices changes and changes in psycho-behavioral and EEG index.

This is the first clinical trial combining tDCS with rTMS for the treatment of schizophrenia patients with predominantly negative symptoms. This study will provide solid evidence for the combination of tDCS with rTMS for the treatment of negative symptoms in schizophrenia. This study will also help to further explore the mechanisms of tDCS combined with rTMS for the treatment of negative symptoms in schizophrenia in terms of imaging and behavior.

DETAILED DESCRIPTION:
This study was designed as an interventional, double-blind, sham-controlled, randomized open-label trial. The main objective is to investigate whether tDCS combined with rTMS is effective in improving negative symptoms in patients with schizophrenia and whether it is superior to single physical therapy. We will also study the effects of tDCS combined with rTMS on blood biomarkers, brain imaging, EEG and psycho-behavioral aspects in patients with schizophrenia.

Schizophrenia patients with prominent negative symptoms who met the inclusion criteria were randomly assigned in a 1:1:1:1 ratio to the active tDCS stimulation combined with active rTMS stimulation, active rTMS stimulation combined with sham tDCS stimulation, and active tDCS stimulation combined with sham rTMS stimulation to sham tDCS stimulation combined with sham rTMS stimulation. General information such as age, gender and marital status were matched between the different groups.

Firstly, a well-trained team is involved in the enrollment process, including a senior psychiatrist, two research nurses, two master students working full-time, and 20 psychiatrists who were actively referring patients for scientific research. Secondly, by giving a more elaborate explanation of the study goals, including the pros and cons, to both patients and their guardians they now better understand the background and possible relevance of the study.

The study population will include 120 patients with schizophrenia mainly with negative symptoms recruited from the inpatient departments of Tianjin Anding Hospital. Schizophrenia is diagnosed according to the Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM-5). All patients are stabilized with no changes in their treatment over the past 1 month prior to their inclusion.

For all patients, clinicians assess the subject's eligibility and provide to each subject and to the patient's legal representative comprehensive verbal and written information regarding the objectives and procedures of the study as well as the possible risks. A signed informed consent is obtained from each participant and/or legal representative for schizophrenia prior to undertaking any study-related procedure. Schizophrenia who do not wish to take part in the study will continue to undergo treatment as usual.

Examinations and assessments during treatment include physical examination, scale assessments, medication use inventory, and laboratory examinations. Subjects were not intervened to take medication during this period. Only detailed recordings were performed.

EEG recording and testing procedures were performed using a 64-conductor Ag/AgC1 electrode cap (Easycap, Berlin, Germany) based on the International 10/20 system extension, and EEG signals were recorded using the BrainAmp DC (Brain Products, Germany) EEG system. There are 4 paradigms in EEG recordings, including P50, P300, MMN and Gamma (20/30/40 Hz). Signal processing was performed offline using BrainVision Analyzer 2.2 (Brain Products, Germany) software.

Four paradigms are used in the experiment to explore the responses related to emotions and cognition, namely task-switching, the color Stroop task, the n-back task, and the Taylor aggression paradigm, at baseline and after interventions. The paradigm order is determined by the Latin square design. The presentation of stimuli and recording of responses are controlled by E-Prime 2 software.

Patients undergo two MRI scan sessions, both including T1, BOLD and DTI. The first session takes place before the treatment starts while the second session takes place in week 4. During this procedure, participants will be exposed to a 3 Tesla magnetic field strength with switching gradient fields, radio waves, and scanner noise. An anatomical scan will be made to obtain the structural image necessary for the localization of functional activation. Patients will only be included in the study upon agreeing to be informed of any coincidental pathological findings. A statement to that effect must be signed before entering into the study. A functional MRI scan (either ASL or EPI) is recorded during the resting state, i.e. the subjects do not do any tasks during this scan. Breathing and heart rate are measured in order to remove variance that correlates with these rhythms.

The primary endpoints of all participants were assessed at the beginning (baseline), at the end of 2 weeks (midpoint) and at the end of 4 weeks (endpoint), then at the 2 weeks after intervention (follow-up point). Other visits were conducted between baseline and 6-week to assess secondary endpoints. The first assessment occurred at baseline prior to randomization. The final assessment occurred after the completion of the 2-week follow-up.

Subjects received care as usual while participating in this study and receiving conventional antipsychotic medication. No adjustment of the type or dose of atypical antipsychotic medication during the previous 1 month and the next 1 month. No interference with the drug regimen, just detailed records. Subjects receive the assessments of clinical symptoms and cognitive function during the week before and after treatment, while blood samples and brain imaging data and behavioral indicators data are collected.

ELIGIBILITY:
Inclusion Criteria:

1. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic classification criteria for schizophrenia.
2. Age 18-60 years old, gender is not limited.
3. Predominantly negative symptoms (PANSS-negative symptom score≥20; or PANSS negative scores are higher than positive scores).
4. Stable psychiatric symptoms (negative symptoms, positive symptoms) for more than 4 weeks or more.
5. No adjustment in the type or dose of antipsychotics taken in the past 1 months and in the next 1 months
6. Patients and Guardians agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with severe physical illness, infectious diseases and immune system diseases, severe neurological diseases, mental retardation or organic brain diseases.
2. Pregnant or lactating women.
3. Other brain stimulation treatment (ECT, MECT, etc) within past 3 months.
4. History of previous seizures.
5. Those evaluated as unsuitable for tDCS and rTMS and those who do not cooperate with treatment.

Additional exclusion criteria for patients participating in the MRI scanning Participants have to fill out a detailed questionnaire covering safety aspects in relation to research in a 3 Tesla magnetic field and MRI environment. These criteria are:

1. MRI incompatible implants in the body (such as cochlear implant, insulin pump, pace maker or other metal implants).
2. Any risk of having metal particles in the eye, due to manual work without proper eye protections.
3. Tattoos containing red pigments.
4. Claustrophobia.
5. The refusal to be informed of structural brain abnormalities that could be detected during the experiment.

   -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Scale for Assessment of Negative Symptoms (SANS) | weeks 0, 2, 4, and 6
  The primary clinical outcome was the overall severity of negative symptoms of psychosis, as measured by the Scale for Assessment of Negative Symptoms (SANS) at weeks 0(baseline), 2,4 and 6.
  And the changes between the four assessments were compared in order of time progression。 The Scale for Assessment of Negative Symptoms (SANS) contains 5 subscales, namely: flat or sluggish affect, poor thinking, lack of will, lack of interest or socialization, and attention deficit. The score range is 0-120, and the total score reflects the severity of negative symptoms; the higher the score, the more severe the symptoms.

SECONDARY OUTCOMES:
Changes in the Positive and Negative symptom scale (PANSS) | weeks 0, 2, 4, and 6
  The secondary clinical outcome was the overall severity of psychotic positive and negative symptoms, as measured by the Positive and Negative Symptom Assessment Scale (PANSS) at week 0 (baseline),2,4 and 6.
  The Positive and Negative Symptom Assessment Scale (PANSS) contains three components: a positive subscale, a negative subscale, and a general psychopathology subscale. The positive scale score range is 7-49, the negative scale score range is 7-49, and the general psychopathology subscale score range is 16-112. Positive and negative symptom assessment scales (PANSS) scores range from 30-210; the higher the score, the more severe the psychiatric symptoms.
Changes in brain imaging markers | weeks 0 and 4
  Patients underwent two MRI scans. The first is performed before the start of treatment, while the second is performed at week 4. During this procedure, participants will be exposed to a 3 Tesla magnetic field strength with switching gradient fields, radio waves and scanner noise. Anatomical scans will be performed to obtain images of the structures needed to localize functional activation. Record functional MRI scans (ASL or EPI) during the resting state, i.e. the subject does not perform any task during the scan. Measure respiration and heart rate to eliminate differences associated with these rhythms.
Changes in Event-related potentials markers | weeks 0 and 4
  Electroencephalogram (EEG) recording and testing procedures were performed using a 64-conductor Ag/AgC1 electrode cap (Easycap, Berlin, Germany) based on the International 10/20 system extension and EEG signals were recorded using the BrainAmp DC (Brain Products, Germany) EEG system. Four EEG signals, P50, P300, MMN and Gamma 20/30/40, were obtained at baseline and post-intervention, respectively. P50 is elicited by a dual-click paradigm. P300 used three stimuli "oddball" evoked paradigms to elicit N1, P2, P3a and P3b ERPs. MMN stimulation used the "oddball" excitation paradigm: Stimuli consisted of 1200 trials presented to the subjects through foam insert earphones. For Gamma 20/30/40 participants were fixated on a computer monitor while listening to up to 500 ms of 20 Hz, 30 Hz and 40 Hz click training of the crosshairs.
Changes in psycho-behavioral markers | weeks 0 and 4
  Four paradigms were used in the experiment to explore responses related to emotion and cognition, i.e., task switching, color tracing task, n-back task, and Taylor attack paradigm, at baseline and after the intervention. The order of the paradigms was determined by the Latin square design. Stimulus presentation and recording of responses were controlled by E-Prime 2 software. Subjects were tested individually and sat at a comfortable viewing distance from the monitor. The experimenter was present in the room throughout the experiment. The experiments all started with a practice area to familiarize the subjects with the content and operation of each task. The experimenter probed the subjects to see if they understood the procedures and clarified instructions when necessary.
MATRICS Consensus Cognitive Battery (MCCB) | weeks 0, 4, and 6
  Cognition
Changes in Gene and Protein markers | weeks 0 and 4
  Blood biomarkers, including GWAS and Metabolomics. In addition, we also evaluate biochemical indexes, such as glucose, lipids, cholesterol, HDL, LDL, thyroid hormones, uric acid.

CONTACTS AND LOCATIONS:
Overall Officials: Shen Li, Doctor, Principal Investigator — Tianjin Anding Hospital
Locations (1):
- Jie Li, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Begemann MJ, Brand BA, Curcic-Blake B, Aleman A, Sommer IE. Efficacy of non-invasive brain stimulation on cognitive functioning in brain disorders: a meta-analysis. Psychol Med. 2020 Nov;50(15):2465-2486. doi: 10.1017/S0033291720003670. Epub 2020 Oct 19. PMID 33070785
- [Background] Gainsford K, Fitzgibbon B, Fitzgerald PB, Hoy KE. Transforming treatments for schizophrenia: Virtual reality, brain stimulation and social cognition. Psychiatry Res. 2020 Jun;288:112974. doi: 10.1016/j.psychres.2020.112974. Epub 2020 Apr 19. PMID 32353694
- [Background] Kennedy NI, Lee WH, Frangou S. Efficacy of non-invasive brain stimulation on the symptom dimensions of schizophrenia: A meta-analysis of randomized controlled trials. Eur Psychiatry. 2018 Mar;49:69-77. doi: 10.1016/j.eurpsy.2017.12.025. Epub 2018 Feb 3. PMID 29413808
- [Background] Mitra S, Mehta UM, Binukumar B, Venkatasubramanian G, Thirthalli J. Statistical power estimation in non-invasive brain stimulation studies and its clinical implications: An exploratory study of the meta-analyses. Asian J Psychiatr. 2019 Aug;44:29-34. doi: 10.1016/j.ajp.2019.07.006. Epub 2019 Jul 5. PMID 31302440
- [Background] Edemann-Callesen H, Winter C, Hadar R. Using cortical non-invasive neuromodulation as a potential preventive treatment in schizophrenia - A review. Brain Stimul. 2021 May-Jun;14(3):643-651. doi: 10.1016/j.brs.2021.03.018. Epub 2021 Apr 2. PMID 33819680
- [Background] Khanna A, Pascual-Leone A, Michel CM, Farzan F. Microstates in resting-state EEG: current status and future directions. Neurosci Biobehav Rev. 2015 Feb;49:105-13. doi: 10.1016/j.neubiorev.2014.12.010. Epub 2014 Dec 17. PMID 25526823
- [Background] Sale MV, Mattingley JB, Zalesky A, Cocchi L. Imaging human brain networks to improve the clinical efficacy of non-invasive brain stimulation. Neurosci Biobehav Rev. 2015 Oct;57:187-98. doi: 10.1016/j.neubiorev.2015.09.010. Epub 2015 Sep 26. PMID 26409343
- [Result] Mally J, Stone TW, Sinko G, Geisz N, Dinya E. Long term follow-up study of non-invasive brain stimulation (NBS) (rTMS and tDCS) in Parkinson's disease (PD). Strong age-dependency in the effect of NBS. Brain Res Bull. 2018 Sep;142:78-87. doi: 10.1016/j.brainresbull.2018.06.014. Epub 2018 Jun 26. PMID 29958911